CLINICAL TRIAL: NCT06856863
Title: Correlation Between Personnality Traits and Ability to Learn Oroesophageal Voice
Acronym: CoPerVOO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RCAPHM25_0002; 2025-A00022-47 (Other: IDRCB)
Record Dates: First submitted 2025-02-26; First posted 2025-03-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Laryngectomy; Total Pharyngo-laryngectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study of personality traits in patients able or unable to learn VOO (Experimental)
  Interventions: Behavioral: Test of personality : questionnary

INTERVENTIONS:
Behavioral: Test of personality : questionnary — The questionnary Temperament and Character Inventory (TCI) describes personality through temperament traits governed by the individual's neurobiological systems and predetermined by heredity; and character traits shaped by social and cognitive experience

SUMMARY:
After total laryngectomy and loss of laryngeal phonation, the oro-oesophageal voice (VOO) is a communication option for the patient. It involves little financial outlay and, when mastered, ensures functional communication, but requires time-consuming speech therapy. VOO acquisition depends on a number of factors, including the patient's physiology, personality and socio-cultural environment. Several authors have suggested the influence of psychology on failure to learn VOO, but the studies found in the literature are old and did not use personality tests to objectivize this link through quantitative analysis. Today, the Temperament and Character Inventory (TCI-125) is a personality test used clinically and in research, and appreciated for the quantitative scores it provides.

The aim of our study is to ascertain whether salient personality traits (as measured by the TCI) are common to patients who succeed in learning VOO, compared with those who do not.

40 subjects who underwent total laryngectomy and had access to speech therapy will be included in this study. A speech assessment with audio recording will be performed and acoustic measurements will be taken. Subjects will also take the TCI-125. Finally, a perceptual evaluation by a jury of experts will categorize the subjects as good or poor speakers.

Inclusion period: 24 months Duration of subject participation: 1 day Total duration: 36 months

ELIGIBILITY:
Inclusion Criteria:

* Men or women over 18 years of age
* French-speaking patients
* MoCA score ≥ 16/30
* Patients who have undergone laryngectomy or total pharyngo-laryngectomy between 6 months and 5 years of age
* Patients who have agreed to learn VOO
* Patients who began speech therapy to learn VOO no more than five years ago
* Patients who have had access to speech therapy to learn VOO for at least six months (completed or ongoing)
* Patients who have received information about the study and have not expressed their opposition
* Patients who are beneficiaries of or entitled to social security coverage

Exclusion Criteria:

* Patients who underwent a laryngectomy or total pharyngolaryngectomy more than 5 years ago
* Patients who did not receive speech therapy to learn OVO postoperatively, or who received less than 6 months of therapy
* Patients with a related condition that prevents them from learning VOO (anatomical or physiological abnormality, esophageal stenosis)
* Patients with a related condition that may be responsible for speech or fluency disorders (developmental, organic, or functional speech and language disorders, stuttering, stammering, fluency disorders, neurological speech disorders)
* Patients with uncorrected hearing loss
* Patients unable to receive informed consent about the ongoing research due to impaired psychological or physical health
* MoCA score <16/30
* Patients with definite depressive symptoms (HAD-D score ≥ 11)
* Patients in a period of exclusion from another research protocol at the time of collection of the non-opposition.
* Subjects covered by articles L1121-5 to 1121-8 of the French Public Health Code (minors, adults under guardianship or trusteeship, patients deprived of their liberty, pregnant or breast-feeding women, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-10-14 (Actual); Primary Completion 2027-10-14 (Estimated); Study Completion 2028-10-14 (Estimated)

PRIMARY OUTCOMES:
TCI-defined personality traits in patients able to learn VOO and those unable to learn VOO | From enrollement to the end of the study at 36 months

SECONDARY OUTCOMES:
Comparison of the sub-scores of the 7 dimensions of the TCI questionnaire | From enrollment to the end of the study at 36 months
Measurement of VOO quality (cepstral peak proeminence in dB) from audio recordings between the two groups (able and unable the learn VOO) | From enrollment to the end of the study at 36 months
Measurement of speech rate (in syllables/second) | From enrollment to the end of the study at 36 months
Measurement of articulatory speed (in syllables / seconds excluding pauses) | From enrollment to the end of the study at 36 months

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France